CLINICAL TRIAL: NCT04682821
Title: The Research of Artificial Intelligence Assistance System Effectiveness for Novice Endoscopists Gastroscopy Training
Brief Title: The Research of AI Assistant Gastroscope Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Renmin Hospital of Wuhan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: EA-19-003-19
Record Dates: First submitted 2020-12-20; First posted 2020-12-24 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2020-12

CONDITIONS: Gastroscopy; Training; Artificial Intelligence

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- with Artificial intelligence assistant system (Experimental): The experiment group would receive the training with the help of artificial intelligence assistant system in addition to the common training. The system is an non-invasive AI system which could help the endoscopists to diagnosis and monitor the blind spot during the gastroscope.
  Interventions: Other: Artificial intelligence assistant system
- without Artificial intelligence assistant system (No Intervention): The control group would receive the training without the help of artificial intelligence assistant system. That is, they would receive the common training process.

INTERVENTIONS:
Other: Artificial intelligence assistant system — The intervention is the use of the artificial intelligence assistant system in addition to the common training. The system is an non-invasive AI system which could help the endoscopists to diagnosis and monitor the blind spot during the gastroscope.
  Arms: with Artificial intelligence assistant system

SUMMARY:
In this study, we proposed a prospective study about the effectiveness of artificial intelligence system for gastroscope training in novice endoscopists. The subjects would be divided into two groups. The experimental group would be trained in painless gastroscopy with the assistance of the artificial intelligence assistant system. The artificial intelligence assistant system can prompt abnormal lesions and the parts covered by the examination (the stomach is divided into 26 parts). The control group would receive routine painless gastroscopy training without special prompts. Then we compare the gastroscopy operation score, coverage rate of blind spots in gastroscopy,check the average test score before and after training, training satisfaction, detection rate of lesions and so on between the two group.

DETAILED DESCRIPTION:
In this study, we proposed a prospective study about the effectiveness of artificial intelligence system for gastroscope training in novice endoscopists. The subjects would be divided into two groups. The experimental group would be trained in painless gastroscopy with the assistance of the artificial intelligence assistant system. The artificial intelligence assistant system can prompt abnormal lesions and the parts covered by the examination (the stomach is divided into 26 parts). The control group would receive routine painless gastroscopy training without special prompts. Then we compare the gastroscopy operation score, coverage rate of blind spots in gastroscopy,check the average test score before and after training, training satisfaction, detection rate of lesions and so on between the two group.

ELIGIBILITY:
Novice endoscopists：

Inclusion Criteria:

1. Males or females who are over 18 years old;
2. After qualified medical education and obtained the Certificate of Chinese medical practitioner;

Exclusion Criterial:

1. A doctor who has already been trained in gastroenteroscopy;
2. Doctors without qualified medical education and didn't obtaine the Certificate of Chinese medical practitioner;
3. The researcher believes that the subjects are not suitable for participating in clinical trials.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 288 (Actual)
Dates: Start 2020-12-23 (Actual); Primary Completion 2021-05-25 (Actual); Study Completion 2021-06-26 (Actual)

PRIMARY OUTCOMES:
Gastroscopy operation score | three month
  Using a professional gastroscopy operation scoring scale, the full score is 100 points, and the score is divided into small items. In this experiment, the effect of training between the two groups was compared by comparing the scores of gastroscopy operation in the experimental group and the control group.

SECONDARY OUTCOMES:
Coverage rate of blind spots in gastroscopy | three month
  Evaluate the gastroscope operation videos retained by each physician during the examination, and calculate the coverage of 26 parts of the gastric mucosa in the experimental group and the control group during the examination. The calculation method is: the coverage rate of the blind area of the gastroscopy = the actual number of parts covered by the examination/26 parts of the stomach x 100%.
Check the average test score before and after training | three month
  the difference between the theoretical test score after the training and the theoretical test score before the training, the calculation method: the theoretical test score after the training-the theoretical test score before the training.
Training satisfaction | three month
  An AI assistant group fills out a questionnaire after training, and determines the satisfaction with AI assistant training through a grading method.
Detection rate of lesions | three month
  the detection rate of lesions in the experimental group and the control group by gastroscopy. Calculation method = number of gastroscopes with detected lesions/total number of gastroscopes completed by beginner physicians x 100%.

CONTACTS AND LOCATIONS:
Overall Officials: Honggang W Yu, Doctor, Principal Investigator — Renmin Hospital of Wuhan University
Locations (1):
- Renmin Hospital of Wuhan University, Wuhan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huang L, Liu J, Wu L, Xu M, Yao L, Zhang L, Shang R, Zhang M, Xiong Q, Wang D, Dong Z, Xu Y, Li J, Zhu Y, Gong D, Wu H, Yu H. Impact of Computer-Assisted System on the Learning Curve and Quality in Esophagogastroduodenoscopy: Randomized Controlled Trial. Front Med (Lausanne). 2021 Dec 14;8:781256. doi: 10.3389/fmed.2021.781256. eCollection 2021. PMID 34970565